CLINICAL TRIAL: NCT02066545
Title: A Phase 2, Randomized, Vehicle-Controlled, Double-Blind, Multicenter Study to Evaluate the Safety and Efficacy of Three Once-Daily CLS001 Topical Gels Versus Vehicle Administered for 12 Weeks to Subjects With Acne Vulgaris
Brief Title: Safety and Efficacy Study of CLS001Topical Gel Compared to Vehicle in Subjects With Inflammatory Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-003
Record Dates: First submitted 2014-02-18; First posted 2014-02-19 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Vehicle Gel (Placebo Comparator)
  Interventions: Drug: CLS001 Topical Gel Vehicle
- CLS001 topical gel 1% (Experimental): Topical application once daily
  Interventions: Drug: CLS001 Topical Gel
- CLS001 topical gel 1.75% (Experimental): Topical application once daily
  Interventions: Drug: CLS001 Topical Gel
- CLS001 topical gel 2.5% (Experimental): Topical application once daily
  Interventions: Drug: CLS001 Topical Gel

INTERVENTIONS:
Drug: CLS001 Topical Gel
  Arms: CLS001 topical gel 1%; CLS001 topical gel 1.75%; CLS001 topical gel 2.5%
Drug: CLS001 Topical Gel Vehicle
  Arms: Vehicle Gel

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of once-daily topical application of CLS001 1%, 1.75% and 2.5% topical gel compared to vehicle topical gel in subjects with inflammatory acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects with facial acne vulgaris, 12 years of age or older.
* Subjects with ≥20 inflammatory facial lesions (papules, pustules) inclusive of the nose, with a maximum of 9 inflammatory pustules.
* An Investigator's Global Assessment (IGA) of Moderate (3) or Severe (4)

Exclusion Criteria:

* Subjects with acne conglobate, acne fulminans, and secondary acne (chloracne, drug-induced acne, polycystic ovarian syndrome, etc.)
* Subjects with greater that 75 facial non-inflammatory lesions (open and/or closed comedones; excluding the nose)
* Subjects with more than 2 facial nodulocystic lesions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion count from Baseline | 6, 9 and 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline at each visit in inflammatory lesions, non-inflammatory lesions and total lesions | 1, 3, 6, 9 and 12 weeks
Absolute change from Baseline at each visit in inflammatory lesions, no-inflammatory lesions, and total lesions | 1, 3, 6, 9 and 12 weeks
Percentage of subjects with an Investigator's Global Assessment (IGA) of clear or almost clear (0 or 1) at each visit | 1, 3, 6, 9, and 12 weeks
Percentage of subjects with a 2 grade reduction in the IGA at each visit | 1, 3, 6, 9, and 12 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Encino Research Center, Encino, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Skin Care Research, Inc., Boca Raton, Florida
  - Belleair Research Center, Pinellas Park, Florida
  - Moore Clinical Research, Inc., Tampa, Florida
  - Kenneth R. Beer, MD, PA, West Palm Beach, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Manhattan Dermatology & Cosmetic Center, New York, New York
  - Derm Research Center of New York, Inc., Stony Brook, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Premier Research, Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Premier Clinical Research, Spokane, Washington